CLINICAL TRIAL: NCT01431027
Title: Left Ventricular Torsional Hysteresis: A Global Parameter for Diastolic Function
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: F101215002; 5R01HL104018 (NIH)
Record Dates: First submitted 2011-08-03; First posted 2011-09-09 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure; Diastolic Heart Failure; Heart Failure With Normal Ejection Fraction
Keywords: Heart Failure; Diastolic Heart Failure; Heart Failure with Normal Ejection Fraction
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diastolic Function: Patients scheduled for cardiac catheterization.

SUMMARY:
Diastolic dysfunction refers to abnormal mechanical properties of the myocardium and includes abnormal LV diastolic distensibility, impaired filling and slow or delayed relaxation- regardless of whether the ejection fraction is normal or depressed and whether the patient is asymptomatic or symptomatic. Epidemiologic studies have demonstrated high prevalence of diastolic heart failure (DHF). The quality of life of these patients is impaired and the clinical outcomes are similar to those with heart failure with systolic dysfunction. Therefore diastolic dysfunction has significant adverse economic impact that is expected to grow further with time. Clinical characteristics alone may not be sufficient to diagnose diastolic dysfunction. A number of invasive and non-invasive parameters have been proposed to diagnose diastolic dysfunction. Most of the presently used non-invasive parameters have a number of limitations. High fidelity measurement of the left ventricular pressures is needed to accurately diagnose diastolic dysfunction. Obtaining it in routine clinical practice is impractical.

In this protocol the investigators have proposed a novel non-invasive parameter called 'Torsional Hysteresis' as a measure of diastolic function. This will be measured using non-invasive cardiac MRI technique. During left ventricular contraction and relaxation, myocardium deforms. During cardiac cycle the myocardium goes back to baseline state prior to beginning of each contraction. However the rate with which it returns to the baseline state is variable. Torsion indicates relative wringing motion of the ventricle around a left ventricular axis and is a global parameter of left ventricular deformation. The parameters have defined a new parameter called torsional hysteresis based on non invasive cardiac MRI assessment. The parameters have hypothesized that for diastolic dysfunction, the torsional hysteresis area is increased as compared to no diastolic dysfunction group.

ELIGIBILITY:
Inclusion Criteria:

Major inclusion criteria: Normal screening LV ejection fraction.

Exclusion Criteria:

1. Atrial fibrillation or other significant cardiac arrhythmia on ECG
2. Presence of pacemaker or defibrillator
3. Angioplasty or primary coronary intervention PCI/PTCA during index cardiac catheterization.
4. Patient is unable to undergo cardiac MRI due to contraindication to MRI (MRI incompatible metal prosthesis or implants or significant claustrophobia).
5. Patient taking phosphodiesterase 5 inhibitor (eg. sildenafil) will be excluded due to potential interaction with nitroglycerin.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To show that torsional hysteresis relates to invasive hemodynamic measure of diastolic function | one time at enrollment
  To show that torsional hysteresis relates to invasive hemodynamic measure of diastolic function: a) Exponential fall of pressure during isovolumic relaxation phase by the time constant of relaxation, tau and b) LV end diastolic pressure-volume relationship (EDPVR).

SECONDARY OUTCOMES:
To demonstrate that torsional hysteresis is a relatively load independent measure of global diastolic function | one time at enrollment
  To demonstrate that torsional hysteresis is a relatively load independent measure of global diastolic function by evaluating effects of nitroglycerin (NTG) on torsional hysteresis and correlating it to invasive hemodynamic measure of diastolic function including a) tau and b) EDPVR.
To evaluate the sensitivity and specificity of torsional hysteresis in diagnosing diastolic dysfunction | one time at enrollment
  To evaluate the sensitivity and specificity of torsional hysteresis in diagnosing diastolic dysfunction (as defined by invasive hemodynamic parameters: tau, EDPVR) and compare it to echocardiographic tissue Doppler assessment in patients undergoing cardiac catheterization for suspected diastolic dysfunction

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VA Medical Center, Birmingham, Alabama
  - UAB Hospital, Birmingham, Alabama